CLINICAL TRIAL: NCT01272817
Title: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation Using Antithymocyte Globulin With Either Melphalan and Cladribine or Total Lymphoid Irradiation
Brief Title: Nonmyeloablative Allogeneic Transplant
Acronym: Mini-allo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#13-6255
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria; Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma; Multiple Myeloma; Waldenstrom Macroglobulinemia; Breast Cancer; Renal Cell Carcinoma; Melanoma; Sarcoma; Ovarian Cancer; Thymoma
Keywords: Nonmyeloablative transplant; Allogeneic transplant; Transplant
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia; Breast Neoplasms; Carcinoma, Renal Cell; Melanoma; Sarcoma; Ovarian Neoplasms; Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cladribine + melphalan (Other): Cladribine + melphalan conditioning
  Interventions: Procedure: Nonmyeloablative Allogeneic Transplant
- TLI (Other): Total lymphoid irradiation conditioning
  Interventions: Procedure: Nonmyeloablative Allogeneic Transplant

INTERVENTIONS:
Procedure: Nonmyeloablative Allogeneic Transplant — Cladribine 0.14 mg/kg/day for five days, melphalan 100 mg/m2 on one day
  Arms: Cladribine + melphalan
Procedure: Nonmyeloablative Allogeneic Transplant — Total lymphoid irradiation 100cGy/day times 10 days (Monday through Friday)
  Arms: TLI

SUMMARY:
Allogeneic transplant from a matched sibling for the treatment of a variety of illnesses including bone marrow failure states, leukemias, myelodysplastic or myeloproliferative syndromes, lymphoma, or myeloma using a nonmyeloablative preparative regimen.

DETAILED DESCRIPTION:
same

ELIGIBILITY:
Inclusion Criteria:

1. Age > 55 years or
2. Age < 55 and LVEF < 45% or creatinine clearance < 60 ml/min
3. Ability to cover the cost of the transplant, necessary medications, and transportation/housing.
4. Caregiver must be available while outpatient

Guidelines for Cladribine-Melphalan-based conditioning:

* Bone Marrow Failure States Severe Aplastic Anemia (relapsed following immunosuppressive therapy) Paroxysmal Nocturnal Hemoglobinuria (poor prognostic features or hemosiderosis)
* AML (first CR except for t(15;17), inv16, t(8,21); second CR; relapse failing second induction attempt)
* ALL (first CR with at least one poor prognostic feature; second or greater CR; relapse failing reinduction attempt)
* MDS (RAEB, RAEBiT, CMMoL)
* CML (chronic phase; accelerated phase; blast phase following reinduction attempt; 2nd chronic or accelerated phase following gleevec therapy
* Hodgkin's lymphoma (first or greater relapse)
* Non-Hodgkin's Lymphoma
* Aggressive Histology (includes T Cell NHL) Incomplete response to induction Second CR Sensitive or refractory relapse
* Indolent Histology Second or greater relapse
* Mantle Cell Lymphoma (any Stage - must have received induction chemotherapy)
* Multiple Myeloma (10% residual plasmacytosis following anthracycline-based chemotherapy or residual disease following autologous transplant)
* Waldenstrom Macroglobulinemia (must have failed either purine analogue-based chemotherapy (Fludara or 2CdA) or standard CVP therapy; hyperviscosity or cytopenias)

Guidelines for total lymphoid irradiation-based conditioning

* MDS (RA, RARS)
* CLL (Rai stage III or IV - must have received at least two different treatment regimens in the past)
* Breast Cancer (symptomatic metastatic disease, who have failed standard chemotherapy)
* Renal Cell Cancer (metastatic disease at multiple sites)
* Malignant Melanoma (metastatic disease at multiple sites)
* Sarcoma (all subtypes presently, unresectable metastatic disease)
* Ovarian Cancer (stage III or IV, platinum insensitive disease, i.e. progression within 6 months of initial platinum chemotherapy)
* Thymoma (unresectable disease)

Exclusion Criteria:

1. Prior allogeneic stem cell or bone marrow transplant
2. Current or past history of invasive mycotic infection
3. Breast Feeding

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Engraftment | One year
  Evaluation of engraftment of donor stem cells by bone marrow examinations at days 30, 100, and 360 after transplant.

SECONDARY OUTCOMES:
Graft-versus-host disease | One year
  Assess the incidence and severity of acute and/or chronic GVHD for patients transplanted on this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Andrey, M.D., Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States